CLINICAL TRIAL: NCT01801332
Title: Intensive Enteral Nutrition in Association With Corticosteroids in Severe Acute Alcoholic Hepatitis: a Multicenter, Randomized, Controlled Trial
Brief Title: Intensive Enteral Nutrition and Acute Alcoholic Hepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Christophe MORENO, Clinical director of the liver unit, Department of Gastroenterology, Hepatopancreatology and Digestive oncology, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NETI HAA
Record Dates: First submitted 2013-02-27; First posted 2013-02-28 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Severe Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intensive arm (Experimental): Corticosteroïds (Methylprednisolone 32 mg/d) for 28 days + intensive enteral nutrition by feeding tube for 14 days
  Interventions: Dietary Supplement: intensive nutrition
- control arm (Active Comparator): Corticosteroïds (Methylprednisolone 32 mg/d) for 28 days + " classical " oral alimentation for 14 days
  Interventions: Dietary Supplement: usual meals

INTERVENTIONS:
Dietary Supplement: intensive nutrition — Patients randomized in " intensive enteral nutrition " arm will receive by feeding tube (with the use of a microsonde), and in continuous administration, 2 liters of Fresubin HP Energy (1500 kcal/liter, 75 gr prot/liter) for patients with a weight of more than 90 kgs (after ascites removal), 1.5 liters of Fresubin HP Energy for patients with a weight between 60 and 90 kgs, and 1 liter of Fresubin HP Energy for patients of less than 60 kgs. Patients with significant encephalopathy despite therapy against encephalopathy will receive Fresubin Hepa in place of Fresubin HP Energy (1300 kcal/liter, 40 gr prot/liter, 44 % branched AA). Duration of enteral nutrition by feeding tube will be 14 days. The adaptation to the targeted volume must be achieved in maximum 3 days. Enteral nutrition will be administered by nasogastric microsonde.
  Arms: intensive arm
Dietary Supplement: usual meals — Patients randomized in " classical oral nutrition " arm (control arm) will receive usual meals (estimated at 1750 kcal/day; 70 g protein/day), and alimentary supplements between meals to achieve the ESPEN recommandations (35-40 kcal/kg/day; protein 1.2-1.5 g/kg/day) (Plauth et al, Clinical Nutrition 2006). Calories and proteins intake must be recorded daily.
  Arms: control arm

SUMMARY:
To evaluate the effect of an intensive enteral nutrition (compared to clinical routine) in association with corticosteroïds in patients with severe acute alcoholic hepatitis.

DETAILED DESCRIPTION:
Acute alcoholic hepatitis (AAH) is characterized by hepatocellular necrosis, ballooning degeneration and an inflammatory reaction with many polymorphonuclear leukocytes, and fibrosis (Mezey E. Treatment of alcoholic liver disease. Semin Liver Dis 1993). The presence of a severe AAH was identified by the presence of a discriminant function (DF) ≥ 32. DF ≥ 32 has been shown to prospectively identify patients with a 40 to 50 % risk of dying within 2 months (Ramond et al, NEJM 1992). The main treatment of AAH consists of abstinence from alcohol. Corticosteroids are generally recommended in patients with severe AAH. Indeed, a recent analysis of the individual data of the patients from the last three randomized controlled trials showed a significantly higher 1-month survival in corticosteroids compared to placebo treated patients with a severe AAH (Mathurin et al, J hepatol 2002). However, efficacy of this therapy is insufficient, since around 40 % of patients with a severe AAH do not respond to corticosteroids (Louvet et al, Hepatology 2007). Moreover, corticosteroïds are still contraindicated in case of active infection or gastrointestinal bleeding, which are relatively common complications in those patients. Therefore, alternative therapeutic options are needed and must be a medical priority.

Alcoholic patients with severe AAH are frequently malnourished and usually remain anorectic for several weeks (DiCecco SR et al, Nutr Clin Pract 2006). Some data indicate that malnutrition is a factor of bad prognosis in this disease. Recent evidence was also provided that adequate enteral nutritional support might have an important impact on long-term survival in those patients (Cabré et al, Hepatology 2000). However, up to now, no study evaluated potential synergetic effect of intensive enteral nutrition and corticosteroids. Moreover, in clinical practice, in the majority of the centers, patients with alcoholic hepatitis receive alimentary supplements and dietetic counseling, which is often insufficient and difficult to apply and to follow.

Aim :

To evaluate the effect of an intensive enteral nutrition (compared to clinical routine which consists in oral supplements) in association with corticosteroïds in patients with severe acute alcoholic hepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Acute alcoholic hepatitis proven by a liver biopsy (necessary histological findings : neutrophils infiltration, ballooned hepatocytes and Mallory bodies)
* Presence of a severe disease, defined by a Maddrey score higher than or equal to 32, at screening and in baseline (day 0). Maddrey score = total bilirubin in mg/dl + 4,6 X (Prothrombin time patient in sec - prothrombin time control in sec)
* Age between 18 and 75 years old, extremes included
* Recent jaundice or in recent aggravation (less than 3 months)
* Chronic alcohol consumption (more than 40 g/day)
* Informed consent read, understand and signed by the patient (in case of significant encephalopathy, a family representative can signed in place of the patient)
* Maximal delay between admission and randomization of 14 days.

Exclusion Criteria:

* Other disease compromising 6 months survival of the patient
* Positive HIV or HCV serology, positive HBs Antigen
* Uncontrolled bacterial or fungal infection (infection must be judged controlled for at least 3 days)
* Uncontrolled upper GI bleeding (bleeding must be controlled for at least 5 days)
* Type 1 Hepatorenal syndrome (creatinin upper than 2,5 mg/dl), as defined by Salerno F et al, Gut 2007;56:1310-1318
* History of bariatric surgery
* Pentoxyphilline therapy
* MARS therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
survival | 6 months survival

SECONDARY OUTCOMES:
survival | 1 month

OTHER OUTCOMES:
infection rate during hospitalisation, early bilirubin change (day 7), Lille score, development of hepatorenal syndrome | entire study duration (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Moreno, MD, PhD, Principal Investigator — Erasme University Hospital
Locations (19):
- Belgium (17):
  - UZ Antwerpen, Antwerp
  - AZ Brugge, Bruges
  - CHU Saint-Pierre, Brussels
  - CHU Brugmann, Brussels
  - Erasme University Hospital, Brussels
  - AZ VUB, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Hôpitaux Iris-Sud, Brussels
  - UZ Gent, Ghent
  - Hôpital de Jolimont, La Louvière
  - KU Leuven, Leuven
  - CHR La Citadelle, Liège
  - Hôpital Saint-Joseph, Liège
  - ULG Sart Tilman, Liège
  - CHR Saint Joseph-Warquignies, Mons
  - Hôpital Ambroise Paré, Mons
  - Hôpital Ottignies, Ottignies-Louvain-la-Neuve
- France (2):
  - CHU Caen, Caen
  - CHU Lille, Lille

REFERENCES:
- [Derived] Moreno C, Deltenre P, Senterre C, Louvet A, Gustot T, Bastens B, Hittelet A, Piquet MA, Laleman W, Orlent H, Lasser L, Serste T, Starkel P, De Koninck X, Negrin Dastis S, Delwaide J, Colle I, de Galocsy C, Francque S, Langlet P, Putzeys V, Reynaert H, Degre D, Trepo E. Intensive Enteral Nutrition Is Ineffective for Patients With Severe Alcoholic Hepatitis Treated With Corticosteroids. Gastroenterology. 2016 Apr;150(4):903-10.e8. doi: 10.1053/j.gastro.2015.12.038. Epub 2016 Jan 5. PMID 26764182